CLINICAL TRIAL: NCT00035867
Title: Phase 1-2a Study of TLK199 HCl Liposomes for Injection in Myelodysplastic Syndrome
Brief Title: Study of TLK199 HCl Liposomes for Injection in Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK199.1001
Record Dates: First submitted 2002-05-06; First posted 2002-05-07 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2005-06

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Injections

INTERVENTIONS:
Drug: TLK199 HCl Liposomes for Injection

SUMMARY:
The purpose of this study is to determine the safety and efficacy of TLK199 in patients with myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of MDS
* Adequate liver and kidney function
* Ineligible for, or refusing, allogeneic bone marrow transplant
* At least 18 years of age
* Discontinuation of growth factors (e.g., G- CSF) at least 2 weeks prior to study entry

Exclusion Criteria:

* Failure to recover from any prior surgery, or any major surgery within 4 weeks of study entry
* Pregnant or lactating women
* History of allergy to eggs
* Other investigational drugs within 14 days of study entry
* Chemotherapy, radiotherapy or immunotherapy within 14 days of study entry
* Concomitant steroids or hormones for the treatment of neoplasms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2002-04; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Oregon Health & Science University, Portland, Oregon
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Cancer Associates, Dallas, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Raza A, Galili N, Callander N, Ochoa L, Piro L, Emanuel P, Williams S, Burris H 3rd, Faderl S, Estrov Z, Curtin P, Larson RA, Keck JG, Jones M, Meng L, Brown GL. Phase 1-2a multicenter dose-escalation study of ezatiostat hydrochloride liposomes for injection (Telintra, TLK199), a novel glutathione analog prodrug in patients with myelodysplastic syndrome. J Hematol Oncol. 2009 May 13;2:20. doi: 10.1186/1756-8722-2-20. PMID 19439093